CLINICAL TRIAL: NCT00805038
Title: Transplant Navigator Intervention to Overcome Barriers to Kidney Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB07-00301
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Results first posted 2011-07-15 (Estimated); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): Usual care
  Interventions: Behavioral: Usual care
- Intervention (Experimental): Navigator will assist patients in completing steps in transplant process
  Interventions: Behavioral: Transplant navigator

INTERVENTIONS:
Behavioral: Transplant navigator — Navigator will provide help to patients in completing specific steps in transplant process.
  Other Names: Control: usual care
  Arms: Intervention
Behavioral: Usual care — Nephrologists and dialysis facilities will provide usual care regarding access to transplantation.
  Arms: Control

SUMMARY:
Compared with chronic dialysis treatment, kidney transplantation generally offers a longer life span, a better quality of life, and lower health care costs for the over 500,000 Americans with End Stage Renal Disease. Despite Medicare funding of virtually all kidney transplants, minority, female, and poor patients with End Stage Renal Disease have decreased access to kidney transplantation. In prior work, the investigators identified the steps in the transplant process that are responsible for creating these disparities. These include medical suitability, interest in receiving a transplant, referral to a transplant center for a pre-transplant workup, placement on a waiting list or identification of a living donor, and receipt of a kidney from a deceased or living donor. The investigators now propose to train transplant recipients to act as transplant navigators and then test the value of using transplant navigators to help patients and providers complete these steps.

The proposed community-based randomized controlled trial will involve approximately 75-100 adult hemodialysis patients at intervention dialysis facilities and approximately 75-100 patients at control facilities to compare a transplant navigator intervention with usual care over a 24 month interval. Baseline evaluation will include sociodemographic and medical characteristics, specific steps completed in the transplant process, and barriers to moving forward in the transplant process. At periodic intervals, the navigator will provide tailored information and assistance to patients and their nephrologists to help them complete the tasks required at each step. The major outcome will be completion of additional steps in the transplant process. Secondary analyses will examine impediments to successful intervention among subjects who fail to move forward in the transplant process despite assistance from a navigator.

The proposed project will test a novel intervention that targets patients and nephrologists as they together make transplant-related decisions. Future work will involve determining the impact of navigators on disparities in transplant rates, examining the cost-effectiveness of transplant navigators, and disseminating the intervention for use across the country. Helping patients complete steps in the transplant process may lead not only to improved access to kidney transplantation but also to better patient survival, decreased health care costs, and increased quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old
* English speaking
* Mentally competent

Exclusion Criteria:

* Prior pre-transplant workup
* Prior kidney transplant
* Active systemic infection
* Active or recent malignancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2009-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ash Sehgal, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Campbell ZC, Dawson JK, Kirkendall SM, McCaffery KJ, Jansen J, Campbell KL, Lee VW, Webster AC. Interventions for improving health literacy in people with chronic kidney disease. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD012026. doi: 10.1002/14651858.CD012026.pub2. PMID 36472416

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: Usual care received by participants
- Transplant Navigator: Navigator will assist patients in completing steps in transplant process
Period: Overall Study
Arm/Group | Usual Care | Transplant Navigator
Started | 75 | 92
Completed | 75 | 92
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Transplant Navigator | Total
Number analyzed (Participants) | 75 | 92 | 167
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 84 | 141
  >=65 years | 18 | 8 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (9) | 54 (10) | 56 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 45 | 73
  Male | 47 | 47 | 94
Region of Enrollment [Number; unit: participants]
  United States | 75 | 92 | 167

OUTCOME MEASURES:

1. Primary Outcome: Number of Steps Completed in Transplant Process
Description: Many kidney failure patients, particularly minorities and women, face barriers in completing the steps required to obtain a transplant. These sequential steps include: medical suitability, interest in transplant, referral to a transplant center, first visit to center, transplant workup, successful candidate, waiting list or identify living donor, and receive transplant. We calculated the number of transplant process steps completed by both groups.
Time Frame: 18-24 months
Population: ITT analysis. Last observation carried forward for preliminary analyses.
Measure: Mean (95% Confidence Interval); unit: steps per participant
Arm/Group | Usual Care | Transplant Navigator
Number analyzed (Participants) | 75 | 92
steps per participant | 1.0 [0.6 to 1.4] | 2.8 [2.4 to 3.2]

2. Secondary Outcome: Impediments to Successful Intervention
Time Frame: 18-24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Usual Care | Transplant Navigator
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/92
Other Adverse Events (participants affected / at risk) | 0/75 | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No